CLINICAL TRIAL: NCT00991640
Title: Impact of an Integrated Obesity Management System on Patient's Care
Acronym: ROGMF-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Marie-France Langlois, Pincipal investigator, Université de Sherbrooke
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 09-022
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention
- Preceptorships (Experimental): Preceptorships with e-learning
  Interventions: Behavioral: 2-day preceptorship on obesity management

INTERVENTIONS:
Behavioral: 2-day preceptorship on obesity management
  Arms: Preceptorships

SUMMARY:
The investigators developed a program aimed at enhancing primary care physician (PCP) teams' expertise, self-efficacy and attitudes with respect to obesity management. The investigators implemented and evaluated this obesity management system based on a preceptorship combined with a virtual learning community favouring continuous support of family medicine groups (FMGs, Groupes de Médecine Familiale) by a team of experts in obesity management; significant improvements regarding their attitudes and perception of self-efficacy were observed immediately after the preceptorship and maintained after one year. Furthermore, the investigators observed significant changes in their practice that were maintained one year later.

The investigators hypothesize that their program combining preceptorships with a virtual community will improve: (1) management and weight loss of obese/overweight subjects who are treated by PCPs for hypertension (HTN), type 2 diabetes (DM2) or impaired glucose tolerance (IGT); and (2) screening and initial management of obesity among unselected patients of PCPs who practice in FMGs.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have, during the past 2 years, at least 4 documented visits for the targeted diseases group and at least 2 visits for the regular follow-up group

Exclusion Criteria:

* Active mental health problem
* Active psychiatric disorder
* Cancer in the last five years
* Patient with medication that changed in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Among patients from the targeted diseases group, we aim at improving: a)the proportion of subjects who have an initial intervention planned, according to the CCPGO; b)the proportion of subjects who lose at least 5% of their initial weight. | 18 months
Among patients from the regular follow-up group, we aim at improving: a)the proportion of patients who have measured weight, BMI and waist circumference and b)the proportion of overweight or obese subjects who have an initial intervention planned. | 18 months

SECONDARY OUTCOMES:
Among health professionals who receive the intervention (vs. those who did not), we aim at ameliorating their attitudes and perceptions towards patients and treatment effectiveness. | 12 months
Among health professionals who receive the intervention (vs. those who did not), we aim at improving their perception of self-efficacy in managing obesity. | 12 months
Among health professionals who receive the intervention (vs. those who did not), we aim at increasing their knowledge and expertise on obesity management and changing their practice. | 12 months
Among patients who are followed by PCPs who receive the intervention (vs. no intervention), we aim at:a) evaluating their attitudes and perceptions regarding obesity/overweight and lifestyle and b)improving their satisfaction regarding their management. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada

REFERENCES:
- [Derived] Baillargeon JP, St-Cyr-Tribble D, Xhignesse M, Grant A, Brown C, Langlois MF. Impact of an integrated obesity management system on patient's care - research protocol. BMC Obes. 2014 Sep 3;1:19. doi: 10.1186/s40608-014-0019-z. eCollection 2014. PMID 26217506